CLINICAL TRIAL: NCT05160909
Title: The Effects of Surgical Positioning on Arthroscopic Shoulder Stabilization: A Prospective Comparison
Brief Title: Evaluation of Surgical Positioning in Arthroscopic Shoulder Stabilization
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Other Study IDs: MBis21E.593
Record Dates: First submitted 2021-12-06; First posted 2021-12-16 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Shoulder Dislocation
MeSH Terms: conditions — Shoulder Dislocation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Beach Chair: Patient positioned in beach chair position during arthroscopic shoulder stabilization
  Interventions: Procedure: Beach Chair Position
- Lateral decubitus: Patient positioned in lateral decubitus position during arthroscopic shoulder stabilization
  Interventions: Procedure: Lateral Decubitus Position

INTERVENTIONS:
Procedure: Beach Chair Position — Patients positioned in beach chair during arthroscopic shoulder stabilization
  Groups: Beach Chair
Procedure: Lateral Decubitus Position — Patients positioned in lateral decubitus position during arthroscopic shoulder stabilization
  Groups: Lateral decubitus

SUMMARY:
The purpose of this study is to prospectively determine whether intra-operative factors, complications and post-operative outcomes differ between beach chair and lateral decubitus surgical positioning for patients receiving arthroscopic shoulder stabilization (anterior or posterior) due to shoulder instability.

ELIGIBILITY:
Inclusion Criteria:

-Any patient undergoing arthroscopic labral repair due to shoulder instability, with or without concomitant debridement.

Exclusion Criteria:

* Revision stabilization surgery
* No previous Bankart repairs, labral repairs, capsulorrhaphy, or Latarjet
* Multidirectional shoulder instability
* Concomitant rotator cuff repair, biceps tenodesis/tenotomy, HAGL repair
* Isolated SLAP repair/labral repair in association with mechanism other than -instability (eg: overhead athletes) open procedures for instability

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who undergo arthroscopic labral repair due to shoulder instability, with or without concomitant debridement.
Sampling Method: Non-Probability Sample
Enrollment: 556 (Estimated)
Dates: Start 2021-12-06 (Actual); Primary Completion 2023-12-06 (Estimated); Study Completion 2023-12-06 (Estimated)

PRIMARY OUTCOMES:
Shoulder instability | 2 years
  Participants will be asked by their surgeon at routine follow up visits if they have encountered any episodes of shoulder instability (shoulder dislocations)

SECONDARY OUTCOMES:
Postoperative patient satisfaction | 2 years
  Participant satisfaction will be measured using the American Shoulder and Elbow Surgeons score (ASES)
Postoperative patient satisfaction | 2 years
  Participant satisfaction will be measured using the Single Assessment Numerical Evaluation survey (SANE)
Postoperative patient satisfaction | 2 years
  Participant satisfaction will be measured using the Western Ontario Shoulder Instability (WOSI) index

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Orthopaedic Institute, Philadelphia, Pennsylvania, United States